CLINICAL TRIAL: NCT00648193
Title: Single-Dose Fasting Bioequivalence Study of Paroxetine Hydrochloride Tablets (40 mg; Mylan) and Paxil® Tablets (40 mg; GSK) in Healthy Adult Volunteers
Brief Title: Fasting Study of Paroxetine Hydrochloride Tablets 40 mg and Paxil® Tablets 40 mg
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PARO-0678
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Paroxetine; Tablets

ARMS (2):
- 1 (Experimental): Paroxetine hydrochloride 40 mg tablet
  Interventions: Drug: Paroxetine hydrochloride 40 mg tablet
- 2 (Active Comparator): Paxil® 40 mg Table
  Interventions: Drug: Paxil® 40 mg Table

INTERVENTIONS:
Drug: Paroxetine hydrochloride 40 mg tablet — 40mg, single dose fasting
  Arms: 1
Drug: Paxil® 40 mg Table — 40mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study is to investigate the bioequivalence of Mylan's paroxetine hydrochloride 40 mg tablets to GSK's Paxil® 40 mg tablets following a single, oral 40 mg (1 x 40 mg) dose administered under fasting conditions to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and/or female of non-childbearing potential.

   1. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

      1. postmenopausal with an absence of menses for at least one (1) year, or
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy and an absence of bleeding for at least three months
   2. During the course of the study, from study screen until study exit - including the washout period, all men must use a spermicide containing barrier method of contraception (i.e. a condom containing spermicide). This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women with all subjects having a Body Mass Index (BMI) less than or equal to 30 but greater than or equal to 19 (see Part II, Administrative Aspects of Bioequivalence Protocols).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, Hepatitis B and Hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco-containing products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   4. Use of monoamine oxidase inhibitors (MAOIs), pimozide, or thioridazine within 30 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, Hepatitis B, or Hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to paroxetine or any related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
11. History of depression, mania, seizure, akathisia, narrow angle glaucoma, and/or suicidal ideation or behavior (suicidality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Czarnik, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html